CLINICAL TRIAL: NCT01195870
Title: Assessment of Patient Use of a New Device: RebiSmart
Status: Completed | Type: Observational
Sponsor: Merck KGaA, Darmstadt, Germany (Industry)
Collaborators: Merck Serono Limited, UK (Industry)
Responsible Party: Sponsor
Other Study IDs: EMR701068-514
Record Dates: First submitted 2010-08-31; First posted 2010-09-06 (Estimated); Last update posted 2014-02-17 (Estimated); Status verified 2014-02

CONDITIONS: Multiple Sclerosis
Keywords: Multiple sclerosis; Rebif; Interferon beta-1a
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Multiple sclerosis (MS) is a chronic disease which causes inflammation and destruction of the nerves in within the brain and the spinal cord. This disease is one of the most common causes of disability in young adults. A ''relapse'' is a phenomenon that occurs when there is an acute attack of disability as a result of an acute attack on the nervous system. There is usually some degree of recovery after a relapse.

Rebif is licensed in the United Kingdom for the treatment of relapsing MS and is given 3 times a week by injections under the skin. The RebiSmart device is a new injection device which has been developed to help patients with injecting their Rebif treatment.

Currently, all treatments for MS are injectable and require long term patient commitment. Patient compliance to treatment is important for the therapy to work effectively and decrease the risk of relapse episodes. Using a device that makes it easy for patients to inject may potentially improve compliance to treatment and therefore potentially have an impact on the number of relapses patients experience. The RebiSmart device has been developed for patients to inject conveniently and in comfort. The device allows the patient to control certain parameters such as needle depth, needle speed, injection time etc, and also has extra features designed to ease the injection process, such as a dose history calendar and an on-screen injection guide. The aim of this study is to determine what percentage of patients liked using the RebiSmart device and found it ''easy'' or ''very easy'' to use. The study will also determine which of the device features were most useful to the patients.

ELIGIBILITY:
Inclusion Criteria:

* Have relapsing remitting multiple sclerosis
* Between 18 to 65 years old inclusive
* Have been prescribed Rebif for the first time but not yet started treatment
* Rebismart as chosen device
* Be under review by MS nurse
* Having given written informed consent to participate in the study

Exclusion Criteria:

* Injections of Rebif given by someone other than the patient
* Patients unable to use the Rebismart device due to visual or physical impairment
* Patients unwilling to give informed consent
* Contra-indications to Rebif as defined in the Summary of Product Characteristics (SPC).
* Allergy to the antipyretic analgesics that will be advised as prophylaxis for flu-like symptoms

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients, who are under regular review by a Multiple Sclerosis nurse, with relapsing remitting multiple sclerosis who have been prescribed Rebif and have chosen to use the RebiSmart device for drug administration.
Sampling Method: Non-Probability Sample
Enrollment: 63 (Actual)
Dates: Start 2009-07; Primary Completion 2010-09 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
Percentage of subjects who liked using the RebiSmart device based on a score of 6 or more on a Visual Analogue Scale (VAS) at the end of 12-week treatment period | up to week 16

SECONDARY OUTCOMES:
Percentage of patients who found RebiSmart easy or very easy to use at the end of 12-week treatment period | up to week 16
Top three functions of the device patients found most useful; top ranked from 1 to 10 | up to week 16

CONTACTS AND LOCATIONS:
Overall Officials: Dr Gillian L Shepherd, MD, MRCP, Study Director — Merck Serono Limited, UK

REFERENCES:
- [Result] D'Arcy C, Thomas D, Stoneman D, Parkes L. Patient assessment of an electronic device for subcutaneous self-injection of interferon beta-1a for multiple sclerosis: an observational study in the UK and Ireland. Patient Prefer Adherence. 2012;6:55-61. doi: 10.2147/PPA.S26250. Epub 2012 Jan 18. PMID 22298944